CLINICAL TRIAL: NCT03721107
Title: A Phase II Randomized, Double Blind, Placebo-controlled, Parallel Group, Multicenter Study to Evaluate the Safety and Efficacy of Repeated Oral Doses of Blautix in Adult Subjects With Irritable Bowel Syndrome (IBS) Subtypes IBS-C and IBS-D
Brief Title: A Trial for New Treatment of Adult Participants With Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 4D pharma plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BHT-II-002
Record Dates: First submitted 2018-10-01; First posted 2018-10-26 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Irritable Bowel Syndrome
Keywords: constipation; diarrhea
MeSH Terms: conditions — Irritable Bowel Syndrome; Constipation; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind trial design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort C: Blautix (Experimental): Participants diagnosed with Irritable bowel syndrome subtype C (IBS-C) received two capsules of Blautix orally, twice daily for 8 weeks. Maximum daily dose of Blautix (strain of Blautia hydrogenotrophica) will be 10^10 to10^11 most probable number (MPN).
  Interventions: Biological: Blautix
- Cohort C: Placebo (Placebo Comparator): Participants diagnosed with IBS-C received two capsules of placebo matched to Blautix orally, twice daily for 8 weeks.
  Interventions: Other: Placebo
- Cohort D: Blautix (Experimental): Participants diagnosed with Irritable bowel syndrome subtype D (IBS-D) received two capsules of Blautix orally, twice daily for 8 weeks. Maximum daily dose of Blautix (strain of Blautia hydrogenotrophica) will be 10^10 to10^11 MPN.
  Interventions: Biological: Blautix
- Cohort D Placebo (Placebo Comparator): Participants diagnosed with IBS-D received two capsules of placebo matched to Blautix orally, twice daily for 8 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Blautix — Blautix is a live biotherapeutic product consisting of a lyophilised formulation of a proprietary strain of bacterium. The study dosing regimen was two capsules two times per day for the duration of the treatment period.
  Other Names: MRx1234; Blautia Hydrogenotrophica
  Arms: Cohort C: Blautix; Cohort D: Blautix
Other: Placebo — Placebo control
  Arms: Cohort C: Placebo; Cohort D Placebo

SUMMARY:
A study to evaluate the effectiveness of oral doses of Blautix in adult participants with irritable bowel syndrome (IBS).

DETAILED DESCRIPTION:
Participants with a diagnosis of IBS will be enrolled as defined by Rome IV criteria and will be classified into cohorts according to the Rome IV classification of IBS subtypes.

Each cohort (Cohort C and Cohort D) will recruit participants who will randomly receive either Blautix or matching placebo in a 1:1 ratio overall of treated to control participants.

Participants will undergo five visits in total across approximately 13 weeks. During the study treatment phase, participants will be asked to complete a variety of Quality of Life questionnaires at certain time points. These will consist of abdominal pain intensity score, IBS symptom severity (IBS-SSS), IBS quality of life (IBS-QoL), hospital anxiety and depression score (HADS), stool frequency, stool consistency & food frequency questionnaire.

Participants will be required to produce relevant blood, urine and faecal samples at pre-determined timepoints from screening through to End of Treatment and follow up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent on an Institutional Review Board (IRB)/ Independent Ethics Committee (IEC) approved informed consent form before any study specific evaluation
2. Males and Females between 18 and 70 years of age
3. Body Mass Index (BMI): 18-39 kg/m^2
4. Having IBS-C or IBS-D as defined by Rome IV* including Subtype Classification as defined in Table 2

   * Recurrent abdominal pain on average, at least 1 day/week in the last 3 months associated with two or more of the following criteria:
   * Related to defecation
   * Associated with a change in frequency of stool
   * Associated with a change in form (appearance) of stool
5. Have a moderate or severe IBS symptom severity score (> 175) as defined by IBS-SSS

Table 2:

IBS -C Abdominal Pain Intensity: weekly average of worst daily (in past 24 hours) abdominal pain score of > 3.0 on a 0 to 10-point scale And Stool Frequency: more than 25% of bowel movements with a consistency of Type 1 or Type 2 Bristol stool chart and less than 25% of bowel movements with Bristol stool form Type 6 or Type 7. Participants must have fewer than 3 complete spontaneous bowel movements (CSBMs) within a one week period (7 days)

IBS-D Abdominal Pain Intensity: weekly average of worst daily (in past 24 hours) abdominal pain score of > 3.0 on a 0 to 10-point scale And Stool Consistency: more than 25% of bowel movements with a consistency of Type 6 or Type 7 Bristol stool chart and less than 25% of bowel movements with Bristol stool form Type 1 or Type 2.Participants must have at least one Type 6 or Type 7 bowel movements on at least four days within a one week period (7 days).

Exclusion Criteria:

1. Males or females <18 and >70 years of age
2. Have a IBS symptom severity score < 175 as defined by IBS-SSS
3. BMI: <18 or >39 kg/m^2
4. Have a significant acute or chronic coexisting illness (cardiovascular, gastrointestinal, endocrine, immunological, metabolic or any condition which contraindicates, in the investigators' judgment, entry to the study)
5. Confirmed clinical diagnosis of bile acid malabsorption and / or on medication for bile acid malabsorption
6. Individuals who, in the opinion of the investigator, are poor attendees or unlikely for any reason to be able to comply with the study requirements
7. Participant is currently enrolled in or has not yet completed at least 30 days since ending other investigational device or drug study(s), or participant is receiving other investigational agent(s)
8. Have a malignant disease or any concomitant end-stage organ disease.
9. Females who are pregnant or breast feeding
10. Refusal to use acceptable methods of birth control (true abstinence, sterilisation, birth control pills, injections or contraceptive implants) for fertile participants (females) while on treatment and following completion of 2 menstrual cycles/ months after the last dose of study treatment. For Males, a barrier method of birth control from randomisation until the Follow-Up visit
11. Use of antibiotics within 1 month of screening
12. Use of systemic steroids within the last month
13. Change in dose or introduction of an antipsychotic within the last month
14. Have suffered from a major psychiatric disorder
15. Clinically diagnosed Lactose intolerance
16. Clinically diagnosed Coeliac disease
17. Change of diet e.g. FODMAP, gluten-free within last 3 months
18. Those > 50 will be excluded if their diagnosis of IBS is recent (<12 months) and if they have not had a sigmoidoscopy or colonoscopy within previous 5 years.
19. Any gastrointestinal-related abdominal surgery other than hernia repair or appendectomy
20. Participants taking prucalopride
21. Other investigational procedures while participating in this study are excluded
22. Known HIV infection, or hepatitis A, B, or C active infection
23. Participants with abnormal laboratory values at screening deemed by the investigator to be clinically significant
24. Participants who have taken commercially available probiotics within the last month (30 days prior to randomization)
25. Participants with known or suspected hereditary fructose intolerance, glucose-galactose malabsorption or sucrase-isomaltose insufficiency
26. Participants taking guanylate cyclase agonists, such as linaclotide and lubiprostone

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2020-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eamonn Quigley, Principal Investigator — Houston Methodist Gastroenterology Clinical Research Foundation, Houston, Texas
Locations (34):
- United States (24):
  - Clinical Research Associates, Huntsville, Alabama
  - Elite Clinical Studies, Phoenix, Arizona
  - Translational Research Group, Inc, North Hollywood, California
  - Probe Clinical Research, Riverside, California
  - Connecticut Gastroenterology Clinical Research, Bristol, Connecticut
  - Digestive CARE of North Broward, LLC, Coral Springs, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Orlando Florida BioClinica Research Network, Orlando, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - East Coast Institute for Research, LLC., Saint Augustine, Florida
  - Guardian Angel Research Center, Tampa, Florida
  - Georgia Medical Associates, Snellville, Georgia
  - Evanston Premier Healthcare & Research, LLC., Evanston, Illinois
  - Centex Research, Inc., Lake Charles, Louisiana
  - Capitol Research, Rockville, Maryland
  - Specialists in Gastroenterology, St Louis, Missouri
  - PharmQuest, Greensboro, North Carolina
  - Aventiv Research Inc., Columbus, Ohio
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - WR-ClinSearch, Chattanooga, Tennessee
  - Clinical Neuroscience Solutions, Inc, Memphis, Tennessee
  - Houston Methodist Gastroenterology Associates, Houston, Texas
  - Gulf Coast Medical Research, LLC., Missouri City, Texas
  - Blue Ridge Medical Research, Lynchburg, Virginia
- Cork University Hospital, Cork, Ireland
- United Kingdom (9):
  - MAC Clinical Research (Barnsley), Barnsley
  - MAC Clinical Research (Blackpool), Blackpool
  - MAC Clinical Research (Cannock), Cannock
  - CPS Research, Glasgow
  - MAC Clinical Research (Leeds), Leeds
  - MAC Clinical Research (Liverpool), Liverpool
  - MAC Clinical Research (Manchester), Manchester
  - Wythenshawe Hospital, Manchester
  - MAC Clinical Research (Stockton-on-Tees), Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quigley EMM, Markinson L, Stevenson A, Treasure FP, Lacy BE. Randomised clinical trial: efficacy and safety of the live biotherapeutic product MRx1234 in patients with irritable bowel syndrome. Aliment Pharmacol Ther. 2023 Jan;57(1):81-93. doi: 10.1111/apt.17310. Epub 2022 Nov 11. PMID 36369645

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 366 participants were randomized across 30 study centers in Ireland, United Kingdom, and United States between 11 October 2018 (first participant enrolled) and 13 May 2020 (last participant completed study).
Pre-assignment Details: Participants who met the eligibility criteria were randomized to receive Blautix or Placebo in either Cohort C or Cohort D depending on classification of IBS subtype by the study doctor.
Groups:
- Cohort C: Blautix: Participants diagnosed with Irritable Bowel Syndrome Subtype-C (IBS-C) received two capsules of Blautix orally, twice daily for 8 weeks. Maximum daily dose of Blautix (strain of Blautia hydrogenotrophica) was 10^10 to 10^11 most probable number (MPN).
- Cohort D: Blautix: Participants diagnosed with Irritable Bowel Syndrome Subtype-D (IBS-D) received two capsules of Blautix orally, twice daily for 8 weeks. Maximum daily dose of Blautix (strain of Blautia hydrogenotrophica) was 10^10 to 10^11 MPN.
- Cohort D: Placebo: Participants diagnosed with IBS-D received two capsules of placebo matched to Blautix orally, twice daily for 8 weeks.
Period: Overall Study
Arm/Group | Cohort C: Blautix | Cohort C: Placebo | Cohort D: Blautix | Cohort D: Placebo
Started | 80 | 84 | 98 | 104
Treated | 80 | 84 | 97 | 104
Completed | 75 | 81 | 83 | 92
Not Completed | 5 | 3 | 15 | 12
Not completed — Adverse Event | 1 | 1 | 6 | 5
Not completed — Lost to Follow-up | 2 | 0 | 3 | 0
Not completed — Inclusion/Exclusion Criteria not Met | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 5 | 5
Not completed — Other | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF) included all participants randomized into the study who received at least one dose of Blautix or Placebo.
Groups:
- Cohort C: Blautix: Participants diagnosed with IBS-C received two capsules of Blautix orally, twice daily for 8 weeks. Maximum daily dose of Blautix (strain of Blautia hydrogenotrophica) was 10^10 to 10^11 MPN.
- Cohort D: Blautix: Participants diagnosed with IBS-D received two capsules of Blautix orally, twice daily for 8 weeks. Maximum daily dose of Blautix (strain of Blautia hydrogenotrophica) was 10^10 to 10^11 MPN.
- Total: Total of all reporting groups
Arm/Group | Cohort C: Blautix | Cohort C: Placebo | Cohort D: Blautix | Cohort D: Placebo | Total
Number analyzed (Participants) | 80 | 84 | 97 | 104 | 365
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (13.04) | 45.3 (13.41) | 43.1 (13.65) | 44.9 (14.40) | 44.4 (13.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 69 | 60 | 73 | 269
  Male | 13 | 15 | 37 | 31 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 21 | 10 | 10 | 61
  Not Hispanic or Latino | 60 | 63 | 87 | 94 | 304
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 0 | 2
  Asian | 1 | 0 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 30 | 33 | 7 | 11 | 81
  White | 48 | 50 | 86 | 90 | 274
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Response
Description: Overall responder was a participant who has at least 7 evaluable weeks of data and has reported an improvement in their weekly symptoms (abdominal pain intensity [API] and stool frequency [SF] or consistency [SC]) for greater than or equal to (>=) 50 percent (%) of the treatment period. Improvement for abdominal pain intensity was defined as decrease in weekly average of worst abdominal pain in the past 24 hours score of at least 30% compared with baseline for Cohort C and Cohort D, for stool frequency was defined as increase of 1 or more complete spontaneous bowel movements (CSBM) per week compared with baseline for Cohort C and for stool consistency was defined as decrease at least 50% in the proportion of days per week with at least one stool that has a consistency of Type 6 or 7 compared with baseline for Cohort D. Participants with <4 weeks available were considered non-responders.
Time Frame: Baseline up to Week 8
Population: Full Analysis Set (FAS) included all participants in the safety analysis set who were appropriately randomized into the study. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort C: Blautix | Cohort C: Placebo | Cohort D: Blautix | Cohort D: Placebo
Number analyzed (Participants) | 76 | 82 | 94 | 101
Percentage of Participants | 25.0 | 17.1 | 23.4 | 17.8
Statistical Analysis 1: Comparison: Cohort C: Blautix vs Cohort C: Placebo; Test type: Superiority; p = 0.152, Chi-squared, Corrected — P-value is from a 1-sided Pearson chi-square test with Yates' correction with null hypothesis that the difference in proportions Blautix - placebo <=0 versus the difference is >0. The significance level for rejection of the null hypotheses is 0.10; Difference in Percentage = 7.9, 95% CI 2-sided [-6.0 to 21.9]
Statistical Analysis 2: Comparison: Cohort D: Blautix vs Cohort D: Placebo; Test type: Superiority; p = 0.216, Chi-squared, Corrected — [p-value comment as in outcome 1, analysis 1]; Difference in Percentage = 5.6, 95% CI 2-sided [-6.8 to 18.0]

2. Secondary Outcome: Number of Participants With Treatment-Related Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered study medication and which does not necessarily have a causal relationship with this treatment. A TEAE was defined as an AE that started or worsened in severity on or after the start date of the study treatment and includes all AEs recorded through the follow-up visit. A treatment-related TEAE was a TEAE possibly related to the study treatment.
Time Frame: Baseline up to follow-up visit (up to Week 14)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort C: Blautix | Cohort C: Placebo | Cohort D: Blautix | Cohort D: Placebo
Number analyzed (Participants) | 80 | 84 | 97 | 104
Participants | 5 | 4 | 16 | 14

3. Secondary Outcome: Number of Participants With Response to Subject Global Assessment of Relief
Description: The subject global assessment of relief was collected weekly through the electronic clinical outcome assessment (eCOA) system. It was a comparison of how the participant has felt over the past week with regards to their IBS to the way they felt before entering the study. It was measured on a 5-point Likert scale with the following responses: Completely relieved; considerably relieved; somewhat relieved; unchanged; worse. The total score ranged from 0-20, where higher scores indicated worsening of condition.
Time Frame: Week 1, 4, 8, follow-up visit (Week 12, 13 and 14)
Population: FAS included all participants in the safety analysis set who were appropriately randomized into the study. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "Number analyzed" signifies those participants who were evaluable at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort C: Blautix | Cohort C: Placebo | Cohort D: Blautix | Cohort D: Placebo
Number analyzed (Participants) | 66 | 70 | 84 | 86
Participants
  Week 1: Completely Relieved | 0 | 2 | 2 | 0
  Week 1: Considerably Relieved | 1 | 3 | 1 | 0
  Week 1: Somewhat Relieved | 6 | 6 | 3 | 8
  Week 1: Unchanged | 58 | 56 | 72 | 76
  Week 1: Worse | 1 | 3 | 6 | 2
  Week 4: Completely Relieved: number analyzed (Participants) | 63 | 63 | 73 | 71
  Week 4: Completely Relieved | 1 | 1 | 2 | 1
  Week 4: Considerably Relieved: number analyzed (Participants) | 63 | 63 | 73 | 71
  Week 4: Considerably Relieved | 13 | 7 | 13 | 14
  Week 4: Somewhat Relieved: number analyzed (Participants) | 63 | 63 | 73 | 71
  Week 4: Somewhat Relieved | 31 | 31 | 26 | 24
  Week 4: Unchanged: number analyzed (Participants) | 63 | 63 | 73 | 71
  Week 4: Unchanged | 17 | 19 | 28 | 28
  Week 4: Worse: number analyzed (Participants) | 63 | 63 | 73 | 71
  Week 4: Worse | 1 | 5 | 4 | 4
  Week 8: Completely Relieved: number analyzed (Participants) | 65 | 60 | 68 | 70
  Week 8: Completely Relieved | 2 | 3 | 5 | 3
  Week 8: Considerably Relieved: number analyzed (Participants) | 65 | 60 | 68 | 70
  Week 8: Considerably Relieved | 20 | 13 | 14 | 16
  Week 8: Somewhat Relieved: number analyzed (Participants) | 65 | 60 | 68 | 70
  Week 8: Somewhat Relieved | 24 | 23 | 22 | 26
  Week 8: Unchanged: number analyzed (Participants) | 65 | 60 | 68 | 70
  Week 8: Unchanged | 18 | 19 | 21 | 20
  Week 8: Worse: number analyzed (Participants) | 65 | 60 | 68 | 70
  Week 8: Worse | 1 | 2 | 6 | 5
  Week 12: Completely Relieved: number analyzed (Participants) | 40 | 52 | 50 | 52
  Week 12: Completely Relieved | 5 | 5 | 5 | 2
  Week 12: Considerably Relieved: number analyzed (Participants) | 40 | 52 | 50 | 52
  Week 12: Considerably Relieved | 6 | 11 | 10 | 5
  Week 12: Somewhat Relieved: number analyzed (Participants) | 40 | 52 | 50 | 52
  Week 12: Somewhat Relieved | 13 | 17 | 14 | 16
  Week 12: Unchanged: number analyzed (Participants) | 40 | 52 | 50 | 52
  Week 12: Unchanged | 14 | 16 | 19 | 24
  Week 12: Worse: number analyzed (Participants) | 40 | 52 | 50 | 52
  Week 12: Worse | 2 | 3 | 2 | 5
  Week 13: Completely Relieved: number analyzed (Participants) | 33 | 41 | 40 | 42
  Week 13: Completely Relieved | 4 | 4 | 4 | 3
  Week 13: Considerably Relieved: number analyzed (Participants) | 33 | 41 | 40 | 42
  Week 13: Considerably Relieved | 9 | 12 | 4 | 3
  Week 13: Somewhat Relieved: number analyzed (Participants) | 33 | 41 | 40 | 42
  Week 13: Somewhat Relieved | 12 | 9 | 12 | 14
  Week 13: Unchanged: number analyzed (Participants) | 33 | 41 | 40 | 42
  Week 13: Unchanged | 7 | 12 | 15 | 18
  Week 13: Worse: number analyzed (Participants) | 33 | 41 | 40 | 42
  Week 13: Worse | 1 | 4 | 5 | 4
  Week 14: Completely Relieved: number analyzed (Participants) | 6 | 8 | 11 | 10
  Week 14: Completely Relieved | 2 | 0 | 0 | 1
  Week 14: Considerably Relieved: number analyzed (Participants) | 6 | 8 | 11 | 10
  Week 14: Considerably Relieved | 2 | 2 | 0 | 1
  Week 14: Somewhat Relieved: number analyzed (Participants) | 6 | 8 | 11 | 10
  Week 14: Somewhat Relieved | 2 | 1 | 3 | 1
  Week 14: Unchanged: number analyzed (Participants) | 6 | 8 | 11 | 10
  Week 14: Unchanged | 0 | 5 | 8 | 4
  Week 14: Worse: number analyzed (Participants) | 6 | 8 | 11 | 10
  Week 14: Worse | 0 | 0 | 0 | 3

4. Secondary Outcome: Change in Percentage of Days Per Week With Undesired Stool Consistency From Baseline at Week 1, 4, 8, Follow-up Visit (Week 12, 13 and 14)
Description: Stool consistency of each bowel movement was rated on 7-level Bristol Stool Chart where Type 1 = separate hard lumps, like nuts (hard to pass), Type 2 = sausage-shaped but lumpy, Type 3 = like a sausage but with cracks on the surface, Type 4 = like a sausage or snake, smooth and soft, Type 5 = soft blobs with clear-cut edges (passed easily), Type 6 = fluffy pieces with ragged edges, a mushy stool, Type 7 = watery, no solid pieces; entirely liquid. A score range of 1 to 7 where, 1 or 2 indicates constipation and a score of 6 or 7 indicates diarrhea. Change in percentage of days per week with at least 1 stool with a undesired stool consistency of 1 or 2 for Cohort C and 6 or 7 for Cohort D on the Bristol Stool Chart from baseline at Week 1, 4, 8, Follow-up Visit (Week 12, 13 and 14) was reported.
Time Frame: Baseline, Week 1, 4, 8, follow-up visit (Week 12, 13 and 14)
Population: FAS included all participants in the safety analysis set who were appropriately randomized into the study. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Percentage of days per week
Arm/Group | Cohort C: Blautix | Cohort C: Placebo | Cohort D: Blautix | Cohort D: Placebo
Number analyzed (Participants) | 64 | 73 | 83 | 94
Percentage of days per week
  Change at Week 1 | 0.13 (22.859) | 3.38 (24.412) | -25.67 (28.078) | -23.70 (30.730)
  Change at Week 4: number analyzed (Participants) | 57 | 63 | 74 | 76
  Change at Week 4 | -4.23 (24.470) | -1.99 (24.077) | -32.43 (33.627) | -33.73 (33.615)
  Change at Week 8: number analyzed (Participants) | 53 | 56 | 67 | 70
  Change at Week 8 | -5.93 (26.705) | -0.10 (22.852) | -40.36 (37.595) | -36.91 (35.753)
  Change at Week 12: number analyzed (Participants) | 33 | 46 | 51 | 57
  Change at Week 12 | -5.66 (23.063) | 1.06 (27.027) | -34.09 (41.128) | -42.13 (31.500)
  Change at Week 13: number analyzed (Participants) | 7 | 15 | 17 | 25
  Change at Week 13 | 10.88 (26.517) | -5.16 (19.868) | -29.38 (35.002) | -32.21 (39.679)
  Change at Week 14: number analyzed (Participants) | 2 | 2 | 4 | 6
  Change at Week 14 | -15.48 (1.684) | -2.98 (15.994) | -40.00 (36.216) | -38.10 (36.608)

5. Secondary Outcome: Percent Change From Baseline in Stool Consistency Assessed by Bristol Stool Form Scale (BSFS) at Week 1, 4, 8, Follow-up Visit (Week 12, 13 and 14)
Description: Stool consistency of each bowel movement was assessed by participants using the 7-point BSFS from 1 to 7 where Type 1 = separate hard lumps, like nuts (hard to pass), Type 2 = sausage-shaped but lumpy, Type 3 = like a sausage but with cracks on the surface, Type 4 = like a sausage or snake, smooth and soft, Type 5 = soft blobs with clear-cut edges (passed easily), Type 6 = fluffy pieces with ragged edges, a mushy stool, Type 7 = watery, no solid pieces; entirely liquid. A score of 1 or 2 indicates constipation and a score of 6 or 7 indicates diarrhea. Lower numbers represented more formed stools and higher numbers represented less formed stools. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 1, 4, 8, follow-up visit (Week 12, 13 and 14)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Cohort C: Blautix | Cohort C: Placebo | Cohort D: Blautix | Cohort D: Placebo
Number analyzed (Participants) | 63 | 70 | 83 | 94
Percent Change
  Percent Change at Week 1 | 15.05 (126.940) | 27.65 (129.217) | 32.30 (36.887) | -27.27 (38.590)
  Percent Change at Week 4: number analyzed (Participants) | 57 | 61 | 74 | 76
  Percent Change at Week 4 | -6.36 (122.165) | -7.18 (112.425) | -40.14 (42.757) | -40.60 (40.128)
  Percent Change at Week 8: number analyzed (Participants) | 52 | 54 | 67 | 70
  Percent Change at Week 8 | -12.00 (145.174) | -4.64 (103.202) | -49.32 (45.798) | -42.64 (39.801)
  Percent Change at Week 12: number analyzed (Participants) | 33 | 44 | 51 | 57
  Percent Change at Week 12 | -7.45 (125.537) | 14.75 (144.064) | -36.96 (50.023) | -49.94 (34.638)
  Percent Change at Week 13: number analyzed (Participants) | 7 | 14 | 17 | 25
  Percent Change at Week 13 | 41.07 (143.017) | -40.31 (89.914) | -33.29 (40.067) | -35.91 (44.635)
  Percent Change at Week 14: number analyzed (Participants) | 2 | 2 | 4 | 6
  Percent Change at Week 14 | -100.00 (0.000) | -25.00 (106.066) | -52.50 (49.319) | -43.53 (44.353)

6. Secondary Outcome: Change From Baseline in Weekly Average Stool Frequency Assessed by Bristol Stool Form Scale (BSFS) at Week 1, 4, 8, Follow-up Visit (Week 12, 13 and 14)
Description: Stool frequency was defined as a sum of weekly CSBMs. Participants were reminded to rate all their bowel movements in the Bristol Stool Chart (BSC) before answering the question. Stool types were assessed using the 7-point BSFS where 1 = separate hard lumps, like nuts (hard to pass), 2 = sausage-shaped but lumpy, 3 = like a sausage but with cracks on the surface, 4 = like a sausage or snake, smooth and soft, 5 = soft blobs with clear-cut edges (passed easily), 6 = fluffy pieces with ragged edges, a mushy stool, 7 = watery, no solid pieces; entirely liquid. A score of 1 or 2 indicates constipation and a score of 6 or 7 indicates diarrhea. Weekly stool frequency was based on the daily stool frequency which was calculated as follows: if there was 1 or more entry for BSC, the number of BSC entries was summed up. If on that day laxative was used, the daily stool frequency was set to 0. If an answer to CSBMs, but no BSC entry was provided, the daily stool frequency was set to 0 on that day.
Time Frame: Baseline, Week 1, 4, 8, follow-up visit (Week 12, 13 and 14)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: complete spontaneous bowel movements
Arm/Group | Cohort C: Blautix | Cohort C: Placebo | Cohort D: Blautix | Cohort D: Placebo
Number analyzed (Participants) | 64 | 73 | 83 | 94
complete spontaneous bowel movements
  Change at Week 1 | 1.33 (2.202) | 1.61 (2.416) | -1.07 (2.441) | -1.02 (3.119)
  Change at Week 4: number analyzed (Participants) | 57 | 63 | 74 | 76
  Change at Week 4 | 2.14 (2.348) | 1.87 (2.809) | -1.60 (2.543) | -1.83 (3.389)
  Change at Week 8: number analyzed (Participants) | 53 | 56 | 67 | 70
  Change at Week 8 | 2.00 (2.289) | 2.42 (2.751) | -2.59 (3.012) | -1.97 (3.048)
  Change at Week 12: number analyzed (Participants) | 33 | 46 | 51 | 57
  Change at Week 12 | 1.76 (2.547) | 2.18 (2.762) | -2.29 (2.599) | -2.43 (3.299)
  Change at Week 13: number analyzed (Participants) | 7 | 15 | 17 | 25
  Change at Week 13 | 2.09 (2.489) | 1.98 (2.539) | -2.05 (3.242) | -1.77 (2.804)
  Change at Week 14: number analyzed (Participants) | 2 | 2 | 4 | 6
  Change at Week 14 | 2.56 (0.507) | 1.19 (0.860) | -4.71 (2.626) | -3.54 (4.063)

7. Secondary Outcome: Change From Baseline in IBS Quality of Life (IBS-QOL) Questionnaire Subscale and Total Scores at Week 4, 8 and Follow-up Visit (Weeks 12-14)
Description: Participants were asked to complete a QOL of 34 items which formed 8 scales: dysphoria (8 items), interference with activity (7 items), body image (4 items), health worry (3 items), food avoidance (3 items), social reaction (4 items), sexual (2 items), and relationships (3 items). All 8 scales were rated on a five-point response scale where, 1= not at all, 2= slightly, 3= moderately, 4= quite a bit, 5= extremely or a great deal. Scores for individual items were averaged to obtain a total score for each sub-scale of IBSQoL. Total and subscale scores were transformed to a 0 to 100 point scale (0=lowest score, 100=highest possible score) with higher scores indicating better IBS-specific quality of life. Transformed scale score = (Sum of the items-lowest possible score/Possible raw score range)∗100. A positive change from baseline indicates improved quality of life.
Time Frame: Baseline, Week 4, 8, follow-up visit (Weeks 12-14)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Cohort C: Blautix | Cohort C: Placebo | Cohort D: Blautix | Cohort D: Placebo
Number analyzed (Participants) | 41 | 41 | 47 | 64
Score on a Scale
  Change at Week 4: Total score: number analyzed (Participants) | 41 | 41 | 45 | 64
  Change at Week 4: Total score | 5.67 (16.858) | 5.79 (21.908) | 5.62 (18.087) | 5.93 (13.113)
  Change at Week 4: Dysphoria score: number analyzed (Participants) | 41 | 41 | 45 | 64
  Change at Week 4: Dysphoria score | 5.95 (20.561) | 5.34 (22.881) | 9.17 (22.627) | 5.81 (17.429)
  Change at Week 4: Interference with activity Score: number analyzed (Participants) | 41 | 41 | 45 | 64
  Change at Week 4: Interference with activity Score | 4.79 (16.952) | 6.71 (22.633) | 7.54 (18.230) | 8.26 (16.008)
  Change at Week 4: Body Image Score: number analyzed (Participants) | 41 | 41 | 45 | 64
  Change at Week 4: Body Image Score | 4.88 (23.779) | 7.62 (23.239) | 5.83 (20.703) | 4.10 (17.860)
  Change at Week 4: Health Worry Score: number analyzed (Participants) | 41 | 41 | 45 | 64
  Change at Week 4: Health Worry Score | 10.98 (23.082) | 10.57 (26.940) | 6.85 (19.727) | 7.55 (19.056)
  Change at Week 4: Food Avoidance Score: number analyzed (Participants) | 41 | 41 | 45 | 64
  Change at Week 4: Food Avoidance Score | 6.50 (20.625) | 4.88 (29.461) | 5.56 (19.624) | 7.55 (19.960)
  Change at Week 4: Social Reaction Score: number analyzed (Participants) | 41 | 41 | 45 | 64
  Change at Week 4: Social Reaction Score | 4.12 (16.922) | 2.44 (24.402) | 0.42 (23.963) | 6.64 (14.935)
  Change at Week 4: Sexual Score: number analyzed (Participants) | 41 | 41 | 45 | 64
  Change at Week 4: Sexual Score | 7.32 (29.445) | 1.52 (24.716) | -0.56 (20.288) | 0.39 (19.284)
  Change at Week 4: Relationships Score: number analyzed (Participants) | 41 | 41 | 45 | 64
  Change at Week 4: Relationships Score | 2.85 (21.214) | 5.89 (26.170) | 1.30 (23.500) | 2.73 (17.509)
  Change at Week 8: Total score: number analyzed (Participants) | 38 | 35 | 47 | 53
  Change at Week 8: Total score | 12.27 (20.969) | 8.09 (18.318) | 11.89 (20.933) | 8.37 (18.043)
  Change at Week 8: Dysphoria score: number analyzed (Participants) | 38 | 35 | 47 | 53
  Change at Week 8: Dysphoria score | 13.40 (21.044) | 7.59 (20.085) | 14.23 (26.241) | 12.21 (20.403)
  Change at Week 8: Interference with activity Score: number analyzed (Participants) | 38 | 35 | 47 | 53
  Change at Week 8: Interference with activity Score | 10.15 (26.120) | 10.31 (21.529) | 15.12 (22.944) | 8.96 (20.247)
  Change at Week 8: Body Image Score: number analyzed (Participants) | 38 | 35 | 47 | 53
  Change at Week 8: Body Image Score | 12.83 (22.696) | 8.93 (18.890) | 13.70 (22.217) | 7.43 (23.096)
  Change at Week 8: Health Worry Score: number analyzed (Participants) | 38 | 35 | 47 | 53
  Change at Week 8: Health Worry Score | 17.32 (27.834) | 12.38 (22.810) | 7.80 (22.947) | 7.23 (19.614)
  Change at Week 8: Food Avoidance Score: number analyzed (Participants) | 38 | 35 | 47 | 53
  Change at Week 8: Food Avoidance Score | 17.54 (27.522) | 7.38 (29.412) | 14.01 (22.327) | 6.60 (24.534)
  Change at Week 8: Social Reaction Score: number analyzed (Participants) | 38 | 35 | 47 | 53
  Change at Week 8: Social Reaction Score | 10.69 (21.401) | 3.21 (17.960) | 8.78 (24.473) | 7.55 (20.669)
  Change at Week 8: Sexual Score: number analyzed (Participants) | 38 | 35 | 47 | 53
  Change at Week 8: Sexual Score | 10.53 (24.406) | 3.57 (22.600) | 3.46 (26.797) | 3.30 (26.420)
  Change at Week 8: Relationships Score: number analyzed (Participants) | 38 | 35 | 47 | 53
  Change at Week 8: Relationships Score | 6.36 (19.800) | 9.05 (22.721) | 7.45 (21.858) | 5.35 (20.155)
  Change at Follow-up visit: Total score: number analyzed (Participants) | 34 | 36 | 37 | 38
  Change at Follow-up visit: Total score | 15.55 (21.368) | 8.09 (16.647) | 7.93 (23.919) | 10.80 (19.950)
  Change at Follow-up visit: Dysphoria score: number analyzed (Participants) | 34 | 36 | 37 | 38
  Change at Follow-up visit: Dysphoria score | 15.99 (23.957) | 8.07 (17.236) | 10.47 (30.336) | 11.43 (21.236)
  Change at Follow-up visit: Interference with activity Score: number analyzed (Participants) | 34 | 36 | 37 | 38
  Change at Follow-up visit: Interference with activity Score | 14.50 (23.195) | 12.00 (21.278) | 9.75 (25.417) | 14.94 (26.243)
  Change at Follow-up visit: Body Image Score: number analyzed (Participants) | 34 | 36 | 37 | 38
  Change at Follow-up visit: Body Image Score | 17.10 (21.777) | 9.38 (17.772) | 8.95 (24.409) | 9.38 (25.200)
  Change at Follow-up visit: Health Worry Score: number analyzed (Participants) | 34 | 36 | 37 | 38
  Change at Follow-up visit: Health Worry Score | 19.36 (28.701) | 9.26 (23.382) | 10.14 (23.663) | 14.25 (18.371)
  Change at Follow-up visit: Food Avoidance Score: number analyzed (Participants) | 34 | 36 | 37 | 38
  Change at Follow-up visit: Food Avoidance Score | 16.91 (23.524) | 9.72 (21.776) | 7.43 (24.594) | 9.21 (26.408)
  Change at Follow-up visit: Social Reaction Score: number analyzed (Participants) | 34 | 36 | 37 | 38
  Change at Follow-up visit: Social Reaction Score | 13.79 (24.942) | 1.04 (15.917) | 6.59 (27.676) | 9.38 (23.554)
  Change at Follow-up visit: Sexual Score: number analyzed (Participants) | 34 | 36 | 37 | 38
  Change at Follow-up visit: Sexual Score | 15.07 (26.253) | 3.13 (23.599) | -1.69 (27.507) | 4.93 (25.425)
  Change at Follow-up visit: Relationships Score: number analyzed (Participants) | 34 | 36 | 37 | 38
  Change at Follow-up visit: Relationships Score | 12.25 (22.774) | 7.18 (22.900) | 2.03 (24.799) | 5.26 (22.041)

8. Secondary Outcome: Change From Baseline in IBS Symptom Severity Score (IBS-SSS) at Week 4, 8 and Follow-up Visit (Weeks 12-14)
Description: Participants were asked to complete a questionnaire on the severity of abdominal distension and pain, frequency of abdominal pain, dissatisfaction with bowel habits, and interference of IBS symptoms with daily life. The IBS-SSS was measured on a Visual Analog Scale (VAS scale) in combination with reported numeric values which equated to an overall score. The scale range was from 0 (no symptoms) to 500 (maximum severity). Participants were categorized as having mild (74-174), moderate (175-299), or severe (>300) IBS symptoms based on symptomology. Higher scores were indicative of greater disease severity (worse outcome). A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 4, 8, follow-up visit (Weeks 12-14)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Cohort C: Blautix | Cohort C: Placebo | Cohort D: Blautix | Cohort D: Placebo
Number analyzed (Participants) | 77 | 81 | 83 | 93
Score on a Scale
  Change at Week 4 | -128.87 (143.885) | -141.30 (139.439) | -125.75 (135.258) | -100.97 (114.939)
  Change at Week 8: number analyzed (Participants) | 73 | 79 | 81 | 85
  Change at Week 8 | -168.46 (157.300) | -173.53 (155.253) | -143.55 (143.781) | -133.63 (139.290)
  Change at Follow-up visit: number analyzed (Participants) | 77 | 80 | 83 | 90
  Change at Follow-up visit | -142.49 (149.678) | -160.66 (150.174) | -113.47 (135.064) | -104.76 (146.447)

9. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression (HADS) Total Score at Week 4, 8 and Follow-up Visit (Weeks 12-14)
Description: Participants were asked to complete the HADS which was a 14-item scale (7 items- anxiety and 7 items-depression) that generated ordinal data. Each question was rated on a scale from 0 - 3. The outcome of the HADS questionnaire was two total scores, the HADS-A (for anxiety) and the HADS-D (for depression). Both total scores are graded on a scale of 0 - 21 and can be categorized as Normal (0 - 7), Borderline Abnormal (8 - 10) and Abnormal (11 - 21). Higher scores indicate higher levels of anxiety and depression. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 4, 8, follow-up visit (Weeks 12-14)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Cohort C: Blautix | Cohort C: Placebo | Cohort D: Blautix | Cohort D: Placebo
Number analyzed (Participants) | 41 | 41 | 47 | 64
Score on a Scale
  Change at Week 4: Anxiety total score: number analyzed (Participants) | 41 | 41 | 45 | 64
  Change at Week 4: Anxiety total score | -0.02 (2.612) | 0.22 (2.954) | 0.09 (2.827) | -0.27 (3.243)
  Change at Week 4: Depression total score: number analyzed (Participants) | 41 | 41 | 45 | 64
  Change at Week 4: Depression total score | 0.24 (3.527) | -0.29 (3.303) | 0.22 (2.566) | 0.00 (2.410)
  Change at Week 8: Anxiety total score: number analyzed (Participants) | 38 | 35 | 47 | 53
  Change at Week 8: Anxiety total score | 0.08 (2.981) | -0.09 (3.320) | -0.32 (3.251) | -0.40 (3.213)
  Change at Week 8: Depression total score: number analyzed (Participants) | 38 | 35 | 47 | 53
  Change at Week 8: Depression total score | -0.18 (3.432) | -0.06 (3.556) | 0.19 (2.787) | -0.36 (3.169)
  Change at Follow-up visit: Anxiety total score: number analyzed (Participants) | 34 | 36 | 37 | 38
  Change at Follow-up visit: Anxiety total score | -0.53 (3.360) | 0.06 (2.714) | -0.14 (3.029) | -0.55 (3.375)
  Change at Follow-up visit: Depression total score: number analyzed (Participants) | 34 | 36 | 37 | 38
  Change at Follow-up visit: Depression total score | -0.85 (3.735) | -0.14 (2.939) | 0.51 (3.024) | -0.68 (2.886)

ADVERSE EVENTS:
Time Frame: Baseline up to follow-up visit (up to Week 14)
Description: SAF included all participants randomized into the study who received at least one dose of Blautix or Placebo.
Arm/Group | Cohort C: Blautix | Cohort C: Placebo | Cohort D: Blautix | Cohort D: Placebo
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/84 | 0/97 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/84 | 1/97 | 1/104
Other Adverse Events (participants affected / at risk) | 17/80 | 19/84 | 41/97 | 43/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort C: Blautix (N=80) | Cohort C: Placebo (N=84) | Cohort D: Blautix (N=97) | Cohort D: Placebo (N=104)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort C: Blautix (N=80) | Cohort C: Placebo (N=84) | Cohort D: Blautix (N=97) | Cohort D: Placebo (N=104)
Upper respiratory tract infection (Infections and infestations) | 4 | 3 | 3 | 4
Gastroenteritis (Infections and infestations) | 0 | 1 | 4 | 4
Nasopharyngitis (Infections and infestations) | 2 | 1 | 5 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 1
Vulvovaginal candidiasis (Infections and infestations) | 2 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Lice infestation (Infections and infestations) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral rhinitis (Infections and infestations) | 0 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 5 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 4 | 5
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 3 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0
Early satiety (General disorders) | 0 | 0 | 1 | 0
Thirst (General disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 1
Brachioradial pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/07/NCT03721107/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/07/NCT03721107/SAP_001.pdf